CLINICAL TRIAL: NCT06809972
Title: Synovial Proliferation on Routine Ultrasound: Active or Inactive? A Prospective Study
Brief Title: Synovial Proliferation on Routine Ultrasound: Active or Inactive?
Acronym: 2BEGIN
Status: Not yet recruiting | Type: Observational
Sponsor: Van Creveldkliniek (Other)
Responsible Party: Sponsor-Investigator, Van Creveldkliniek, Center for Benign Hematology, Thrombosis and Haemostasis, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: 2BEGIN
Record Dates: First submitted 2024-10-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Haemophilia; Hemophilia A; Hemophilia B
Keywords: Subclinical synovial proliferation; Ultrasound; MRI; Elastography
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Ultrasound imaging — Ultrasound, MRI and elastography to screen for and follow subclinical synovial changes in ankle, elbow and knee.
  Other Names: MRI; Elastography

SUMMARY:
There is cumulating evidence for the presence of non-observed or subclinical joint bleeding in patients with haemophilia. Early detection of active subclinical synovial proliferation would allow early intervention in order to prevent deterioration of joint health. Patients with subclinical (=non-observed) signs of synovial proliferation in knee(s), ankle(s) and/or elbow(s) will be invited to participate in this study to further characterize the synovial proliferation status (active or inactive) by means of physical examination, MRI, ultrasound and elastography. Synovial proliferation status will be monitored for a maximum period of 12 weeks, during which participants will also receive standard-of-care treatment, i.e. administration of optimized coagulation factor replacement therapy and prescription of the NSAID celecoxib (optional).

DETAILED DESCRIPTION:
To be completed

ELIGIBILITY:
Inclusion Criteria:

* Gender: male
* Patients with severe haemophilia A or B
* Treated with registered prophylaxis medication including coagulation factors and by- passing agents.
* Age ≥ 12 years
* Subclinical synovial proliferation in ≥1 joint (ankle, knee and/or elbow), defined as the presence of hypertrophic synovium, score >0 according to the HEAD-US protocol, as confirmed during routine ultrasound screening.
* Able to give written informed consent.

Exclusion Criteria:

* A major bleed ≤ 3 months or a minor bleed ≤ 1 month prior to inclusion in the joint of interest.
* On demand therapy.
* Currently treated with any type of haemophilia prophylaxis medication.
* Joints with prosthesis or treated with arthrodesis will not be included for physical examination and ultrasound analysis. However, participants may still be included in the study with their other joints.
* Confirmed inflammatory joint diseases such as rheumatoid arthritis or psoriatic arthritis.
* History of inhibitor development (≥ 5 Bethesda Units* (BU) at any time or 1-5 BU for

  * 1 year prior to inclusion.
* Contra-indication for treatment with NSAIDs, (allergy, severe liver failure, renal failure (GFR <30ml/min), congestive heart failure (NYHA II-IV), peripheral arterial disease and/or cerebrovascular disease.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Haemophilia is an X-linked disease.
Study Population: The study population consists of male participants ≥ 12 years of age, with severe haemophilia A or B treated with prophylaxis, who were diagnosed with asymptomatic synovial proliferation in ≥1 joint (ankle, knee and/or elbow) by means of ultrasound imaging during routine screening at the outpatient clinic of the Van Creveldkliniek, UMC Utrecht, the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
- The primary objective of this study is to evaluate the diagnostic accuracy of physical examination and ultrasound to identify active synovial proliferation in haemophilia patients with subclinical synovial hypertrophy. | 12 weeks
  As no gold standard to identify active subclinical proliferation is available, "change in synovial proliferation over time" will be used as surrogate endpoint. This is measured by ultrasound assessment according HEAD-US protocol . Possible outcomes are: no change (baseline HEAD-US score = 12-week follow-up HEAD-US score) or changed (baseline HEAD-US score < or > 12-week follow-up HEAD-US score). Fully recovered synovial proliferation will also be categorized as changed. The diagnostic accuracy will be derived comparing 'change in synovial proliferation' with the 'presumed' definition at baseline (active or inactive).
  Definition of active synovial proliferation at baseline: synovial proliferation on ultrasound and the presence of at least one of the following criteria:
  * HJHS swelling >0
  * Warmth palpation absent/present at baseline
  * JADE Synovial Hyperaemia >0
  * No history of synovial proliferation (yes/no)
  * Hemosiderin on MRI (IPSG>0)
  * Elastography

SECONDARY OUTCOMES:
- To identify predictors for (changes in) synovial proliferation status within participant characteristics (age, baseline treatment, joint bleeding history) and joint characteristics (extent of arthropathy (Pettersson score on X-rays)). | 12 weeks
  Baseline participant characteristics (age, baseline treatment, joint bleeding history) and joint characteristics (extent of arthropathy (Pettersson score on X-rays)) will be extracted from medical files.
- To evaluate the diagnostic accuracy of the presence of synovial hemosiderin, as measured by MRI, to identify active synovial proliferation in haemophilia patients with subclinical synovial hypertrophy. | 12 weeks
  Clinical and ultrasound definition of active synovial proliferation: synovial proliferation on ultrasound (HEAD-US synovium score >0) and the presence of at least one of the following criteria:
  - Hemosiderin on MRI: IPSG score Hemosiderin Deposit > 0 at baseline
- To evaluate the diagnostic accuracy of synovial elastography to identify active synovial proliferation in hemophilia patients with subclinical synovial hypertrophy | 12 weeks
  Clinical and ultrasound definition of active synovial proliferation: synovial proliferation on ultrasound (HEAD-US synovium score >0) and the presence of at least one of the following criteria:
  - Elastography:

OTHER OUTCOMES:
- To describe elastographic differences between active clinical synovitis, active subclinical synovial hypertrophy and inactive subclinical hypertrophy. | At baseline (week 0) without follow-up
  For the side objective a group of patients with active clinical synovitis will only undergo elastography and be used as positive control in elastography-analysis, no other measurement nor analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Lize van Vulpen, MD, PhD, Principal Investigator — University Medical Center Utrecht - Van Creveldkliniek
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Pseudonimyzed data may be shared with other (international) researchers upon request at the principal investigator.
  On group level, data will be presented at congresses and in peer-reviewed articles.
Supporting Information: Analytic Code
Time Frame: 15 years after study closure.
Access Criteria: Please contact the principal investigator, Dr. L.F.D. van Vulpen.